CLINICAL TRIAL: NCT05112757
Title: Effective Conversion of Individuals at Risk
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very low recruitment success and all recruitment options were exhausted
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Collaborators: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICBE-S-000283
Record Dates: First submitted 2021-10-19; First posted 2021-11-09 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Obstructive Sleep Apnea; Atrial Fibrillation
Keywords: OSA; AFib
MeSH Terms: conditions — Sleep Apnea, Obstructive; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Smartphone app use
  Interventions: Other: Smartphone application use

INTERVENTIONS:
Other: Smartphone application use — Use of a smartphone application

SUMMARY:
This study aims to guide participants in recognizing their OSA (obstructive sleep apnea) and AFib (atrial fibrillation) symptoms, realizing what medical conditions can cause these symptoms (if any) and inform the participants on their possible diagnosis

DETAILED DESCRIPTION:
The primary objective is to analyze how many patients at risk of medical conditions will be converted to a health care professional by a smartphone application. Historical data (number of patients at risk of OSA and/or AFib that seeked help for their condition in the past year) from institute will be used as a reference. We will refer to this as the 'baseline conversion rate', reflecting the natural transition of patients in the general healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* High risk of OSA and/or AFib, as defined by the risk algorithm developed by Sanford health
* 18 years or older, with sufficient English language skills
* Owning a smartphone with a relatively new operating system (iOS v. 14 (Iphone 6S or higher) or an Android device v.11<)
* Able to download and handle an app on a smartphone
* Willing and able to give informed consent

Exclusion criteria:

* Diagnosed with OSA and/or AFib
* Diagnosed health issues that are potentially life threatening or causing mental issues (stroke, Alzheimer's Disease, depression, etc.)
* Pregnancy/breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Effective conversion | 6 months after consent
  Number of patients that visited the Primary Care Physician

CONTACTS AND LOCATIONS:
Overall Officials: Tim Weysen, MSc, Principal Investigator — Philips Healthcare
Locations (1):
- Sandford Health, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No